CLINICAL TRIAL: NCT01336842
Title: Phase I Trial of Cisplatin and Pemetrexed in Combination With Panobinostat in Advanced Solid Tumors, With Emphasis on Non-Small Cell Lung Cancer
Brief Title: Study of Cisplatin and Pemetrexed in Combination With Panobinostat in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#220; 222274 (Other: UC Davis); CLBH589BUS31T (Other: Novartis)
Record Dates: First submitted 2011-04-11; First posted 2011-04-18 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Solid Tumors; Non-Small Cell Lung Cancer (NSCLC)
Keywords: panobinostat; cisplatin; pemetrexed; dose escalation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Panobinostat; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase I dose-escalation (Experimental): Drug: panobinostat Drug: cisplatin Drug: pemetrexed Other: Biomarker studies
  Interventions: Drug: Panobinostat, Cisplatin, Pemetrexed

INTERVENTIONS:
Drug: Panobinostat, Cisplatin, Pemetrexed — Drug: Panobinostat Oral (by mouth) once daily every Monday, Wednesday, and Friday for the first two weeks of each three week cycle (as per dose escalation schedule (dose levels 1 and 2: AUC 5; dose levels 3 and 4: AUC 6). Number of cycles: 6 maximum.
  Drug: Cisplatin IV (in the vein) on day 1 of a 21-day cycle Number of cycles: 6 maximum. Drug: Pemetrexed IV (in the vein) on day 1 of a 21-day cycle Other: Correlative studies Biomarker Analysis: blood collected pre-study and Cycles 2-6, Day 1.
  Other Names: LBH-589; Platinol; Almita

SUMMARY:
The purpose of this study is to find out if panobinostat taken with cisplatin and pemetrexed can be used safely without increasing side effects and that the combination will have a better effect than platinum-based doublet chemotherapy alone.

DETAILED DESCRIPTION:
The purpose of this phase I study of oral panobinostat plus cisplatin and pemetrexed is to determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLTs) in patients with advanced solid tumors, with an emphasis in non-small cell lung cancer. Another purpose of this study is to find out if oral panobinostat in combination with cisplatin and pemetrexed can be administered safely without significant increase in toxicity and that the combination will increase efficacy compared to platinum-based doublet chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proven advanced solid tumors for which curative standard treatments are not available.
* Must have measurable or evaluable disease.
* Male or female patients aged ≥ 18 years old.
* Any number of prior chemotherapy regimens.
* ECOG Performance Status of ≤ 2 with a life expectancy greater than 3 months.
* Clinically euthyroid (may be on thyroid hormone replacement)
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of study treatment.
* Ability to provide written informed consent
* Must meet the following laboratory criteria:

Hematology:

* Neutrophil count of ≥ 1.5 x 109/L
* Platelet count of ≥ 100 x 109/L
* Hemoglobin ≥ 9 g/dL

Biochemistry:

* AST/SGOT and ALT/SGPT ≤ 2.5 x upper limit of normal (ULN) or ≤ 5.0 x ULN if the transaminase elevation is due to disease involvement
* Serum bilirubin ≤ 1.5 x ULN
* Serum creatinine ≤ 1.5 x ULN or 24-hour creatinine clearance ≥ 50 ml/min
* Total serum calcium (corrected for serum albumin) or ionized calcium ≥ LLN and ≤ ULN
* Serum potassium ≥ LLN and ≤ ULN
* Serum sodium ≥ LLN and ≤ ULN
* Serum albumin ≥ LLN or 3g/dl
* Serum magnesium ≥ LLN and ≤ ULN
* Any elevated Alkaline Phosphatase due to bone metastasis can be enrolled

Exclusion Criteria:

* Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer.
* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first panobinostat treatment.
* Patients who have received chemotherapy, any investigational drug or undergone major surgery < 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Impaired cardiac function
* Other concurrent severe and/or uncontrolled medical conditions that could cause unacceptable safety risks or compromise compliance with the protocol
* Concomitant use of drugs which are generally recognized to have a risk of causing torsades de pointes where such treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Patients with unresolved diarrhea ≥ CTCAE grade 2
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral panobinostat. Inability to swallow panobinostat capsules whole.
* Concomitant use of any anti-cancer therapy or radiation therapy
* Uncontrolled or symptomatic brain metastases.
* Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not willing to use a double barrier method of contraception during the study and 3 months after the end of treatment. One of these methods of contraception must be a barrier method. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months).
* Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment.
* Known positivity for human immunodeficiency virus (HIV) or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-04; Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility of oral panobinostat in combination with cisplatin and pemetrexed | Within ±3 days of the scheduled day of assessment except for adverse events that will be evaluated continuously through the study. The expected time frame for this outcome measure is 18 weeks (or six cycles)
  Safety assessments will consist of monitoring and recording all adverse events and serious adverse events, the regular monitoring of hematology, blood chemistry and urine values, regular measurement of vital signs and the performance of physical examination. Safety and tolerability will be assessed according to the NCI CTCAE v4.

SECONDARY OUTCOMES:
Maximum-tolerated dose as assessed by NCI CTCAE, Version 4.0 | 3 week cycle; the expected time frame is 18 weeks (or 6 cycles)
  Determination of maximum tolerated dose (MTD) will be based on cycle 1 toxicities
Dose-limiting toxicities and toxicity profile as assessed by NCI CTCAE, Version 4.0 | 3 week cycle; the expected time frame is 18 weeks (or 6 cycles)
  Dose-limiting toxicity (DLT) will be based on cycle 1 toxicities.
Exploratory biomarker analysis | Blood specimens will be collected prior to treatment, prior to Cycles 2-6. In addition, a blood specimen will be collected if the patient is removed from the study due to progression of disease. the expected time frame is 18 weeks (or 6 cycles)
  Molecular markers predictive for response to panobinostat remain unknown. This trial offers the opportunity to retrospectively study biomarkers and their association with clinical outcomes.
Efficacy of oral panobinostat in combination with cisplatin/pemetrexed in an expanded cohort of patients with NSCLC | CT scans will be performed at baseline and every two cycles; the expected time frame is 18 weeks (or 6 cycles)
  Response rate will be assessed by CT scan. CT scans will be performed at baseline and every two cycles. The evaluation of response will be based on standard RECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: David Gandara, MD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - University of California Davis Cancer Center, Sacramento, California
  - Henry Ford Health System, Detroit, Michigan